CLINICAL TRIAL: NCT07232147
Title: Clinical Study on the Safety, Tolerance and Preliminary Efficacy of Human Mesenchymal Stem Cell Therapy for Parkinson's Disease
Brief Title: Clinical Research on Stem Cell Therapy for Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Liaoning Medical Diagnosis and Treatment Technology Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNMDTC
Record Dates: First submitted 2025-08-10; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease (PD); Neurodegenerative Diseases; Movement Disorders
Keywords: Parkinson's disease(PD); Umbilical cord mesenchymal stem cells (hUC-MSCs); Stem cell therapy; Safety and efficacy
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human-derived stromal cells (Experimental): Administer human matrix cells by intravenous infusion or nasal drip once every two weeks, for a total of 5 administrations.
  Interventions: Biological: Human-derived stromal cells

INTERVENTIONS:
Biological: Human-derived stromal cells — The human-derived stromal cells were administered intravenously once every two weeks, for a total of 5 times. Among them, half of the subjects (10 people) received intranasal administration of human-derived stromal cells once a day, in the morning and evening, from the 6th to the 8th day after each administration; the remaining subjects (10 people) received nasal administration of placebo once a day, in the morning and evening, from the 6th to the 8th day after each administration.

SUMMARY:
This study, through different administration methods, adopted a randomized, double-blind, placebo-controlled trial design to evaluate the safety and tolerability of human umbilical cord mesenchymal stem cells (hUC-MSCs) in patients with Parkinson's disease, explore their initial effectiveness and the relationship between biological active factors and therapeutic efficacy. The "Clinical Study on the Treatment of Parkinson's Disease with Human Umbilical Cord Mesenchymal Stem Cells" of this study is expected to provide clinical trial evidence for the development of safe and effective clinical cell therapies for patients with Parkinson's disease.

DETAILED DESCRIPTION:
Research Design and Implementation

(1) Inclusion, Exclusion and Withdrawal Criteria for Participants

1. Case Inclusion Criteria:

   1.1 Male and female individuals aged between 40 and 70 years old, excluding adolescent patients with Parkinson's disease.

   1.2 According to the 2015 MDS Parkinson's disease diagnostic criteria, confirmed by a PI or other movement disorder experts based on medical history, physical examination and neurological examination.

   1.3 Modified Hoehn and Yahr staging under levodopa withdrawal period is less than or equal to 3 levels.

   1.4 Have applied levodopa-like drugs, and have a good response to dopaminergic treatment, that is, compared with the withdrawal period, the UPDRS score (combined Parkinson's disease rating scale) of the subjects during the on period decreased by more than 33%.

   1.5 If the subject is taking any central nervous system acting drugs (such as benzodiazepines, antidepressants, hypnotics), the treatment plan must be optimized and stabilized 90 days before the screening visit.

   1.6 At least 90 days before the screening, stable Parkinson's disease symptom treatment has been carried out, and no additional Parkinson's disease symptom treatment is needed from the baseline visit for at least one year.

   1.7 Pregnant women use reliable contraceptive methods during the period from 30 days before the baseline visit to 6 months after taking the study drug.

   1.8 Participants voluntarily join this study, sign the informed consent form, and fully understand the content, process and possible adverse reactions of the trial, and be able to complete the study according to the requirements of the trial protocol.
2. Case Exclusion Criteria:

   2.1 Atypical or drug-induced Parkinson's disease. 2.2 Any limb UPDRS resting tremor score of 3 or higher. 2.3 Montreal Cognitive Assessment (MoCA) score lower than 25 points. 2.4 Clinical features of psychosis or refractory hallucinations. 2.5 Epilepsy history, and having seizures within the past 6 months. 2.6 Mental retardation, possible or definite suicidal thoughts or behaviors, etc. mental disorders or symptoms.

   2.7 Chronic kidney disease: Glomerular filtration rate (GFR) < 50 ml/min/m2 as the diagnostic criterion.

   2.8 Liver function changes: Alanine transaminase (ALT) > 150 U/L and/or total bilirubin > 1.6 mg/dl.

   2.9 Clinical refractory orthostatic hypotension at the time of screening or at the baseline visit, with a systolic blood pressure change of greater than or equal to 20 mmHg and a diastolic blood pressure change of greater than or equal to 10 mmHg within 2 minutes from a sitting position to standing position, and ineffective with drug treatment or baseline sitting blood pressure less than 90/60 mmHg.

   2.10 Congestive heart failure history, clinically significant bradycardia, second or third degree atrioventricular block.

   2.11 Pulmonary disease: Chronic obstructive pulmonary disease (COPD) or moderate to severe asthma.

   2.12 Active malignant tumors or diagnosed as malignant tumors within 5 years before the screening.

   2.13 Any autoimmune disease or immunodeficiency diagnosis, including recent 3-year chemotherapy or current use of immunosuppressive treatment, white blood cell (WBC) < 3 × 103 cells/ml.

   2.14 Moderate to severe cerebrovascular accident or traumatic brain injury history.

   2.15 Within the past 3 months or planned within the next 6 months to undergo major surgery.

   2.16 Clinically significant abnormalities in the laboratory study during the screening visit.

   2.17 History of using study medication within 30 days before the screening visit.

   2.18 History of brain surgery for Parkinson's disease. 2.19 Unable to return for clinical assessment, laboratory study or imaging assessment during the follow-up.

   2.20 History of drug abuse. 2.21 Active anticoagulation treatment or abnormal INR. 2.22 Other situations that researchers consider would cause significant danger to the subject or complicate the study assessment after enrollment.
3. Withdrawal Criteria: 3.1 If the patient requests to withdraw or if the equivalent dose of levodopa changes by more than 30% compared to the baseline level, the subject is deemed unsuitable to continue the trial.
4. Number of enrolled cases: It is planned to include 20 subjects who meet the inclusion and exclusion criteria.
5. Administration route: Human umbilical cord mesenchymal stem cells were administered via intravenous infusion. Some subjects were also given the treatment through nasal instillation.
6. Administration method: Human umbilical cord mesenchymal stem cells were administered intravenously once every 2 weeks, for a total of 5 times. Among them, half of the subjects (10 people) received nasal instillation of human umbilical cord mesenchymal stem cells once in the morning and once in the evening each day from the 6th to the 8th day after each administration; the remaining subjects (10 people) received nasal instillation of the stem cell solvent (0.9% sodium chloride injection containing 5% human albumin, which is consistent in appearance, packaging, instructions for use, and labels with the nasal administration preparation of human umbilical cord mesenchymal stem cells) once in the morning and once in the evening each day from the 6th to the 8th day after each administration. All subjects should receive basic treatment simultaneously during the trial period.

ELIGIBILITY:
Inclusion Criteria:

The participants must meet all of the following criteria to be included in this study:

1. The participants must fully understand and comply with the research procedures, voluntarily participate in the study and sign the informed consent form;
2. At the time of signing the informed consent, the participants must be aged 18 or above and under 75 years old, with no gender restrictions;
3. During the screening process, the participants must have had primary Parkinson's disease for at least 5 years, have a confirmed medical history record and meet the diagnostic criteria for primary Parkinson's disease as defined by the International Parkinson and Movement Disorder Society (MDS);
4. During the screening, according to the MDS-UPDRS scoring scale, the Hoehn-Yahr classification of the "off" period of drug treatment is 2 to 4;
5. During the screening, the score of the third part of the MDS-UPDRS in the "off" period must be greater than 30;
6. During the screening, the stable duration of Parkinson's disease and the stable duration of the optimized drug dosage must be at least 4 weeks, and the duration of levodopa use must be at least 1 year;
7. During the screening, the participants must have a response to levodopa treatment, and the levodopa loading test must be positive;
8. The participants must experience a decline in the efficacy of anti-Parkinson's disease treatment, which affects their quality of life;
9. The participants must have good compliance and be able to cooperate with the completion of the assessment items of the trial; For participants with reproductive potential and their partners, they must be free from pregnancy plans for at least 2 weeks before the screening to at least 1 year after the administration of the drug, and must agree to take effective non-drug contraceptive measures during the trial (such as condoms, non-drug intrauterine devices, etc.), except for those who have taken permanent contraceptive measures, such as bilateral tubal ligation, vasectomy, etc.

Exclusion Criteria:

If the subjects meet any of the following criteria, they will not be included in this study:

1. Allergic to the study drug or its excipients, or allergic to similar drugs of the study drug, or have a history of severe allergies (including any food allergy or drug allergy);
2. Have a previous history of mental disorders, serious diseases, or other significant diseases that may affect safety;
3. Have a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibody positive), or acquired immunodeficiency syndrome-related diseases, or positive HIV serological test results;
4. Positive for hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCV-Ab), or Treponema pallidum antibody positive;
5. Previously diagnosed with secondary or atypical Parkinson's syndrome caused by drugs, metabolic disorders, or other reasons;
6. Previously diagnosed with epilepsy, stroke, multiple sclerosis, poorly controlled or progressive neurological diseases;
7. Have new or unstable mental symptoms within 1 year before screening (such as mental confusion, severe depression, or tendencies towards self-harm/suicide);
8. Have a history of dementia or severe cognitive dysfunction; or have obvious dementia or cognitive dysfunction at screening; the 1.1 part of the MDS-UPDRS score at screening is > 3; due to dementia, the subject's compliance is affected, diary cannot be accurately recorded, and/or the informed consent cannot be signed;
9. Have other serious systemic diseases at the time of screening;
10. Have any history of malignant tumors in the past;
11. Are participating in other clinical trials, or have participated in other clinical studies within 3 months before administration and received intervention treatment;
12. Have active infections at the screening period, and still need systemic application of antibiotics, antifungal, antiviral treatment at baseline and the infection has not been controlled;
13. Have a history of stroke, unstable angina pectoris, or myocardial infarction attack within 6 months before screening;
14. Have a history of schizophrenia or other severe mental disorders, drug or alcohol abuse;
15. Pregnant or lactating women; Subjects deemed unsuitable for participation in the study by the investigator's comprehensive assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-10 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | From baseline up to 48 weeks
  The safety and tolerability of hUC-MSCs will be assessed by monitoring the frequency of all adverse events (AEs) and serious adverse events (SAEs).
  Measure: Number of participants with AEs and SAEs
Severity of Adverse Events | From baseline up to 48 weeks
  Severity of AEs and SAEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.
  Measure: Grade on NCI-CTCAE v5.0 scale
Safety Assessments: Vital Signs | From baseline up to 48 weeks
  Changes in vital signs including body temperature, heart rate, blood pressure, and oxygen saturation.
  Measure: Number of participants with clinically significant changes in vital signs
Safety Assessments: Laboratory Parameters | From baseline up to 48 weeks
  Changes in laboratory tests including complete blood count, coagulation profile, liver and kidney function, BNP, D-dimer, and serum troponin.
  Measure: Number of participants with clinically significant abnormal laboratory values
Safety Assessments: Physical Examination | From baseline up to 48 weeks
  Findings from physical examinations, including skin lesions/rashes. Measure: Number of participants with clinically significant physical examination findings

SECONDARY OUTCOMES:
Change in Motor Function as Assessed by MDS-UPDRS Part III | Baseline, 4, 16, 28, and 48 weeks
  Change in severity of motor symptoms (e.g., tremor, rigidity, bradykinesia) using the MDS-UPDRS Part III score.
  Measure: Score on MDS-UPDRS Part III
Change in Disease Staging as Assessed by Hoehn & Yahr Staging | Baseline, 4, 16, 28, and 48 weeks
  Change in disease stage using the Hoehn & Yahr Staging scale. Measure: Stage on Hoehn & Yahr scale
Change in Non-Motor Symptoms as Assessed by NMSS | Baseline, 4, 16, 28, and 48 weeks
  Change in non-motor symptoms using the Non-Motor Symptoms Scale (NMSS). Measure: Score on NMSS
Change in Depressive Symptoms as Assessed by HAMD | Baseline, 4, 16, 28, and 48 weeks
  Change in depressive symptoms using the Hamilton Depression Rating Scale (HAMD).
  Measure: Score on HAMD
Change in Anxiety Symptoms as Assessed by HAMA | Baseline, 4, 16, 28, and 48 weeks
  Change in anxiety symptoms using the Hamilton Anxiety Rating Scale (HAMA). Measure: Score on HAMA

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data in this study (including demographic information, baseline characteristics, all efficacy and safety endpoints, imaging assessment data, etc.).
  Related documents: The research plan, statistical analysis plan, informed consent form, and summary of the clinical research report will also be provided.
  Data availability: The data will be made available 6 months after the publication of the primary endpoint results of this study in a peer-reviewed journal, and will be maintained for a period of 5 years.
  Access Conditions: Data access rights will be granted to those researchers who submit proposals for conducting approved, scientifically sound meta-analyses or for other research purposes. Proposals should be sent to [specified email address or data access committee]. Requesters are required to sign a data usage agreement.
  Mechanism: The data will be provided through a controlled-access data warehouse .
Supporting Information: Study Protocol, SAP
Time Frame: Start date: Available within 6 months after the publication of the main results paper of this trial.
  End time: At least 5 days from the date of sharing commencement.
Access Criteria: Data access rights will be granted to those researchers who submit proposals for conducting approved, scientifically sound meta-analyses or for other research purposes. Proposals should be sent to [406083722@@qq.com]. Requesters are required to sign a data usage agreement.